CLINICAL TRIAL: NCT03898141
Title: Animal-assisted Placebo-induced Analgesia: A Randomized Controlled Trial in Healthy Participants
Brief Title: Animal-assisted Placebo-induced Analgesia
Acronym: AAPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: Prof. Undine Lang, University Psychiatric Clinics (UPK), Basel, Switzerland (Unknown)
Responsible Party: Principal Investigator, Dr. Karin Hediger, Principal Investigator, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 006-19-1
Record Dates: First submitted 2019-03-25; First posted 2019-04-01 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Pain; Relations, Researcher-Subject
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled parallel group within-subjects design
Who Masked: Participant
Masking Description: As the employed study design necessitates the deception of participants about the true nature of the used intervention, i.e. placebo cream and the true aim of the dog's presence.
  After the termination of the study, all the subjects are debriefed regarding the real experimental procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Animal-assisted placebo condition (AAPL) (Experimental): Participants will receive verbal information that they are receiving an analgesic cream (i.e. ""Anti-dolor, containing Lidocain "), which has been shown to produce significant pain reduction in previous clinical trials. However, they will receive an inert cream.
  Additionally, they will be told that a dog will be present during the experiment to examine whether animals can be present during experimental studies or if they are too big of a distraction. Prior to the pain assessment, participants are allowed to greet the dog. The intensity of interaction will be documented and be rated on a scale from 1-5 (1=very low degree of interaction, 5=very high de-gree of interaction). During the experiment the dog will be lying in the room with some distance to participants to avoid further physical interaction. The dog will always be lying at the same spot. Therefore, the distance between participant and dog will always be the same. However, partici-pants will still be able to see the dog.
  Interventions: Other: Animal-assisted placebo (AAPL)
- Placebo only (PO) (Placebo Comparator): Participants will receive verbal information that they are receiving an analgesic cream (i.e. ""Anti-dolor, containing Lidocain "), which has been shown to produce significant pain reduction in previous clinical trials. However, they will receive an inert cream.
  Interventions: Other: Placebo (PL)
- Dog only (DO) (Experimental): Participants will be told that a dog will be present during the experiment to examine whether animals can be present during experimental studies or if they are too big of a distraction. Prior to the pain assessment, participants are allowed to greet the dog. The intensity of interaction will be documented and be rated on a scale from 1-5 (1=very low degree of interaction, 5=very high degree of interaction). During the experiment the dog will be lying in the room with some distance to participants to avoid further physical interaction. During the experiment the dog will be lying in the room with some distance to avoid further physical interaction.
  After the introduction of the dog, participant will have the verbal information that the applied cream only moisturizes the skin to allow accurate pain measurements
  Interventions: Other: Dog only (DO)
- No dog, no placebo (ND) (No Intervention): Participants will participant will have the verbal information that the applied cream only moisturizes the skin to allow accurate pain measurements.

INTERVENTIONS:
Other: Placebo (PL) — Participants will get deceptive and receive an inert cream (=placebo intervention) that "reduces pain".
  Arms: Placebo only (PO)
Other: Dog only (DO) — In the dog intervention a dog will be present during the second measurements. However, participants will only learn the true aims of the presence of the dog after the study (delayed informed consent).
  Arms: Dog only (DO)
Other: Animal-assisted placebo (AAPL) — Participants receive the placebo intervention in the presence of a dog.
  Arms: Animal-assisted placebo condition (AAPL)

SUMMARY:
An increased interest of animal-assisted interventions (AAI) can be observed within clinical practice, even though it is still not entirely clear how the presence of an animal contributes to the outcome of a treatment. One theory maintains that the presence of an animal influences the relationship between health-provider and patient, which then in turn affects the outcome of the treatment. To investigate this theory, this study will combine AAI with a placebo intervention, as placebo interventions offer the basic form of intervention working through relationship and expectancy.

The effects of the presence of a dog will be assessed with a standardized experimental heat pain paradigm (TSA-II) in a randomized controlled trial in healthy participants (N=128). After a baseline measurements of heat pain threshold and tolerance, participants will be randomly assigned to one of the following four conditions: a) analgesia-expectation, no dog present, b) analgesia-expectation, dog present, c) no-expectation, no dog present and d) no-expectation, dog present.

The dog will be introduced after randomization. Expectancy will be induced by a deceptive cream which is said to helps against pain. Afterwards, posttreatment measurements will be conducted and participants fill in questionnaires about their perceptions of the experimenter.

DETAILED DESCRIPTION:
Upon arrival, all participants will be asked to read the study information again and sign to confirm their informed consent. They will also be asked to complete the sociodemographic data (SDD) questionnaire.

During the experiment there will be three points of questionnaire-assessment. The following questionnaires will be used: expectancy will be assessed with the Expectancy of Relief Scale. Expectancy of Relief Scale is adapted to the scaling of the primary outcome. Expectancy has been measured in previous studies. It should detect if participants expectancy changes after the intervention phase. Further, it would also be interested to examine if the presence or absence of a dog has an impact on expectancy.

Furthermore, following each pain stimuli participants will be asked to complete two short questions on pain intensity and unpleasantness. Pain intensity and unpleasantness are adapted to the scaling of the primary outcome. Subjective pain intensity and unpleasantness are commonly assessed pain dimensions in heat pain paradigm studies. Intensity entails the cognitive dimensions of pain, whereas unpleasantness comprises the affective dimension of pain. Also, after each pain stimuli participants will complete the Counselor Rating Form-Short (CRF-S) to assess they perception of the experimenter.

After pain measurement, there will be a final assessment, using the credibility and effectiveness of the placebo analgesia expectation (CMQ; adapted Version of the Context Model Questionnaire), as well as the CRF-S and a short questionnaire on participants attitude towards dogs and pets (AAPL questionnaire). Study factors, dependent variables and schedule of the study are represented in Tables 1 and 2.

Before starting with the experimental procedures all participants will be introduced to the TSA-II de-vice and the study procedure. All participants will be assigned to a baseline assessment of heat tolerance and threshold. Participants will be randomized to the four experimental conditions (see below) followed by experimentally induced pain using an established and standardized heat pain paradigm: Heat stimuli will be administered to the right volar forearm using a 30x 30-mm Peltier device (Medoc, Ramatishai, Israel; TSA-II) placed at 2/3 of the distance from wrist to elbow. Heat pain threshold will be determined by the methods of limits. Temperature will be increased from the baseline (32°C) at a rate of 0.5°C /s. Participants are instructed to press the button to determine the turning point from perceiving warmth to the perception of pain. When the pain threshold has been reached, the device will resume from its baseline (32 °C) with a rise of 0.5 °C/s. This procedure will be repeated three times (Locher et al., 2017). Pain threshold will be defined as the average of the three measurements. Pain tolerance will also be determined by the method of limits: Participants will be asked to stop the increasing heat stimulus at the moment they cannot stand the heat any longer. Three measurements will start at 32 °C, with a rise of 0.5 °C/s. Heat tolerance will be defined as the average of the three measurements. Pain threshold will always be measured prior to pain tolerance in order to minimize interference between pain threshold and tolerance. After pain induction, participants will complete in the CMQ and the CRF-S questionnaires to detect how they perceive the experimenter. All instructions will be conveyed in a standardized manner to ensure that the participant-experimenter relationship is comparable in terms of friendliness and attention across all four conditions.

Experimental conditions:

* Placebo condition (PL): Participants will receive verbal information that they are receiving an analgesic cream (i.e. ""Antidolor, containing Lidocain "), which has been shown to produce significant pain reduction in previous clinical trials. However, they will receive an inert cream.
* Animal-assisted placebo condition (AAPL): Participants receive the same verbal information as in the PL condition. Additionally, they will be told that a dog will be present during the experiment to examine whether animals can be present during experimental studies or if they are too big of a distraction. Prior to the pain assessment, participants are allowed to greet the dog. The intensity of interaction will be documented and be rated on a scale from 1-5 (1=very low degree of interaction, 5=very high degree of interaction). During the experiment the dog will be lying in the room with some distance to participants to avoid further physical interaction. The dog will always be lying at the same spot. Therefore, the distance between participant and dog will always be the same. However, participants will still be able to see the dog.
* Dog only condition (DO): Participants will be told that a dog will be present during the experiment to examine whether animals can be present during experimental studies or if they are too big of a distraction. Prior to the pain assessment, participants are allowed to greet the dog. The intensity of interaction will be documented and be rated on a scale from 1-5 (1=very low degree of interaction, 5=very high degree of interaction). During the experiment the dog will be lying in the room with some distance to participants to avoid further physical interaction. During the experiment the dog will be lying in the room with some distance to participants to avoid further physical interaction. The dog will always be lying at the same spot. Therefore, the distance between participant and dog will always be the same. However, participants will still be able to see the dog. After the introduction of the dog, participant will have the verbal information that the applied cream only moisturizes the skin to allow accurate pain measurements.
* No Dog condition (ND): Participants will participant will have the verbal information that the applied cream only moisturizes the skin to allow accurate pain measurements.

After the intervention, pain induction will then be performed for a second time (test phase) and participants complete the CMQ, CRF-S and AAPL questionnaires. Finally, participants will be fully debriefed about the real aims of the experiment (delayed informed consent). The expected study duration will be 70 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Right-handedness

Exclusion Criteria:

* Being scared of dogs or dog hair allergy by self-report
* Any acute or chronic disease (chronic pain, hypertension, heart disease, renal disease, liver disease, diabetes) as well as skin pathologies, neuropathies or nerve entrapment symptoms, sensory abnormalities affecting the tactile or thermal modality
* Current medications (psychoactive medication, narcotics, intake of analgesics) or being currently in psychological or psychiatric treatment
* Insufficient German language skills to understand the instructions
* Previous participation in studies using pain assessment with Peltier Devices
* Current or regular drug consumption (THC, cocaine, heroin, etc.)
* pregnancy
* nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Heat pain tolerance assessed by TSA-II | 30 minutes
  Heat stimuli will be administered to the right volar forearm using a 30x 30-mm Peltier device (Medoc, Ramatishai, Israel; TSA-II) placed at 2/3 of the distance from wrist to elbow. Pain tolerance will be determined by the method of limits: Participants will be asked to stop the increasing heat stimulus at the moment they cannot stand the heat any longer. Three measurements will start at 32 °C, with a rise of 0.5 °C/s. Heat tolerance will be defined as the average of the three measurements.

SECONDARY OUTCOMES:
Participants perception of the experimenter I | 15 minutes
  Participants perception of the experimenter will be conducted via the KMS (Adapted version of the Context Model Questionnaire CMQ) questionnaire twice, after each pain induction phase (baseline and posttreatment).
  KMF has 16 items with a scale from 1-5 (1= not at all, 5= very much, with a higher score indicating a better outcome. All items will be analyzed individual.
Participants perception of the experimenter II | 15 minutes
  Participants perception of the experimenter will also be conducted via the CRF-S questionnaire (Counselor Rating Form Short) twice, after each pain induction phase (baseline and posttreatment).
  CRF-S questions contains 12 items on a scale from 1-7 (1= not much, 7= very much, with a higher score indicating a better outcome. All items will be analyzed individual.
Heat pain threshold assessed by TSA-II | 30 minutes
  Heat pain threshold will be determined by the methods of limits. Temperature will be increased from the baseline (32°C) at a rate of 0.5°C /s. Participants are instructed to press the button to determine the turning point from perceiving warmth to the perception of pain. When the pain threshold has been reached, the device will resume from its baseline (32 °C) with a rise of 0.5 °C/s. This procedure will be repeated three times. Pain threshold will be defined as the average of the three measurements.

OTHER OUTCOMES:
Pain expectancy by the VAS scale (visual analogue scale) | 5 minutes
  This should detect if participants expectancy changes after the intervention phase and if eventually the presence of a dog has an impact on expectancy.
  VAS scale ranges from 0-10 (0 = no pain at all; 10= the worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Division Clinical Psychology and Psychotherapy, Faculty of Psychology, University of Basel, Basel, Base-Stadt, Switzerland

IPD SHARING:
Plan to Share IPD: No
We are planning on sharing the anonymized data on a openly assess platform.

REFERENCES:
- [Background] Hsieh C, Kong J, Kirsch I, Edwards RR, Jensen KB, Kaptchuk TJ, Gollub RL. Well-loved music robustly relieves pain: a randomized, controlled trial. PLoS One. 2014 Sep 11;9(9):e107390. doi: 10.1371/journal.pone.0107390. eCollection 2014. PMID 25211164
- [Background] Locher C, Frey Nascimento A, Kirsch I, Kossowsky J, Meyer A, Gaab J. Is the rationale more important than deception? A randomized controlled trial of open-label placebo analgesia. Pain. 2017 Dec;158(12):2320-2328. doi: 10.1097/j.pain.0000000000001012. PMID 28708766
- [Background] Krummenacher P, Candia V, Folkers G, Schedlowski M, Schonbachler G. Prefrontal cortex modulates placebo analgesia. Pain. 2010 Mar;148(3):368-374. doi: 10.1016/j.pain.2009.09.033. Epub 2009 Oct 28. PMID 19875233
- [Background] Krummenacher P, Kossowsky J, Schwarz C, Brugger P, Kelley JM, Meyer A, Gaab J. Expectancy-induced placebo analgesia in children and the role of magical thinking. J Pain. 2014 Dec;15(12):1282-93. doi: 10.1016/j.jpain.2014.09.005. Epub 2014 Sep 23. PMID 25261340
- [Background] Hermann C, Hohmeister J, Demirakca S, Zohsel K, Flor H. Long-term alteration of pain sensitivity in school-aged children with early pain experiences. Pain. 2006 Dec 5;125(3):278-285. doi: 10.1016/j.pain.2006.08.026. Epub 2006 Oct 2. PMID 17011707
- [Background] Petersen GL, Finnerup NB, Norskov KN, Grosen K, Pilegaard HK, Benedetti F, Price DD, Jensen TS, Vase L. Placebo manipulations reduce hyperalgesia in neuropathic pain. Pain. 2012 Jun;153(6):1292-1300. doi: 10.1016/j.pain.2012.03.011. Epub 2012 Apr 13. PMID 22503337
- [Background] Price DD. Psychological and neural mechanisms of the affective dimension of pain. Science. 2000 Jun 9;288(5472):1769-72. doi: 10.1126/science.288.5472.1769. PMID 10846154
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491